CLINICAL TRIAL: NCT00002082
Title: Azithromycin in the Treatment of Cryptosporidiosis in Patients With Acquired Immune Deficiency Syndrome (AIDS): A Randomized, Multi-Center, Placebo-Controlled, Double-Blind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 058F; 066-143
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Cryptosporidiosis; Acquired Immunodeficiency Syndrome; Azithromycin
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate the safety and efficacy of azithromycin in the treatment of intestinal cryptosporidial infection in AIDS patients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine.
* Antidiarrheal medication with imodium or paregoric only.

Patients must have:

* HIV infection.
* Intestinal cryptosporidiosis proven by stool microscopy on at least two occasions prior to study enrollment.
* Life expectancy of at least 2 weeks by clinical assessment. In states where the legal age of consent for medical procedures is 21 years, patients below the age of 21 must have consent of parent or guardian.

Prior Medication:

Allowed:

* Zidovudine.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known hypersensitivity or significant intolerance to macrolide antibiotics.
* Marked abnormalities of liver or renal function.
* Causes for diarrhea other than, or in addition to, cryptosporidiosis.
* Inability to receive oral medication.

Concurrent Medication:

Excluded:

* Cancer chemotherapy (including therapy for Kaposi's sarcoma).
* Any drug or biologic preparation (e.g., bovine colostrum, paromomycin, spiramycin, somatostatin) with possible anticryptosporidial activity.
* Immunostimulant or lymphocyte replacement therapy.

Prior Medication:

Excluded:

* Another investigational drug within 7 days prior to study enrollment (investigational medications available through a treatment IND will be allowed with the approval of the sponsor, the treatment IND sponsor, and the Pfizer clinical monitor).
* Immunostimulant or lymphocyte replacement therapy.
* Cancer chemotherapy (including therapy for Kaposi's sarcoma).

Not expected to comply with the requirements of the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Infectious Disease Med Group, Oakland, California
  - UCSD Med Ctr, San Diego, California
  - Cornell Univ Med Ctr, New York, New York
  - Univ of Tennessee, Memphis, Tennessee